CLINICAL TRIAL: NCT04752761
Title: Compliance al Rilevamento PROMs Mediante Supporto Digitale e Correlazione Rispetto Alla Rilevazione Ambulatoriale Nella Protesica di Ginocchio
Brief Title: Compliance With PROMs Detection Through Digital Support and Correlation Compared Standard to Outpatient Detection in Knee Prosthetics
Acronym: DIG-PROMs-k
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CE-AVEC 584/2020 / Oss / IOR
Record Dates: First submitted 2020-12-23; First posted 2021-02-12 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Approach-Approach Conflict; Knee Discomfort
Keywords: PROMs; Digital; Knee prosthesis; Oxford knee score

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DIG-PROMs-k (Other): Patients who underwent TKA are given conventional and digital OKS surveys. Patients adhesion to both surveys will be compared.
  Interventions: Behavioral: Extrambulatory digital PROMs detection

INTERVENTIONS:
Behavioral: Extrambulatory digital PROMs detection — An alternative PROMs evaluation method will be used in which the questionnaire will be administered to the patient digitally (Google Forms) in an outpatient environment

SUMMARY:
Two methods for detecting outcomes after knee prosthetic surgery are compared: the traditional one using paper questionnaires administered in the outpatient setting (Oxford Knee Score) VS detection using digital questionnaires created on Google Forms and sent to the patient's smartphone on which the compilation takes place in the extra area outpatient.

DETAILED DESCRIPTION:
PROMs (Patient Reported Outcomes Measures) are used globally for the evaluation of the results of a prosthetic surgery. One of the most used methods in the evaluation of PROMs in knee prosthetic surgery is the Oxford Knee Score, usually measured in an outpatient setting using paper questionnaires.

The aim of the study is to investigate the validity of an alternative method of evaluating PROMs in which the questionnaire will be administered to the patient digitally (Google Forms) in an out-of-patient setting.

The questionnaire aimed at the subjective evaluation of the discomfort induced by arthrosis of the knee (Oxford Knee Score), will be administered during the pre-hospitalization visits and again during the follow-up visits carried out at 1, 3 and 6 months after intervention. The digital evaluation will be sent to the patient during the outpatient visits and will be considered valid only if completed within 48 hours of the same.

On each patient the measurements will be carried out in both methods and differences in terms of compliance and satisfaction with the two methods under examination will be detected. Any differences in the final result of the Oxford Knee Score compared to the two methods and the differences in terms of outpatient assessment times will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients with gonarthrosis with indication of hip arthroplasty
* males and females aged 18-78 and with a Barthel scale score ≥ 91
* patients in possession of private digital electronic support (smartphone, tablet or PC)

Exclusion criteria:

* patients with a Barthel scale score ≤ 90
* patients with psychiatric pathologies, a history of drug and alcohol abuse
* patients not in possession of private digital electronic support

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient's adhesion to the digital Oxford Knee Score compilation after the pre-admission visit | 1 month before surgery (pre-admission outpatient visit)
  Adhesion: The primary end point will be assessed in terms of patient adhesion at the digital survey of the OKS index compared to the conventional one.
  Those who complete the questionnaire within 48 hours of the outpatient visit will be considered as cases with positive adhesion with the digital assessment; those who reply after 48 hours or who do not reply will be considered with negative adhesion.
Patient's adhesion to the digital Oxford Knee Score compilation one month after surgery | 1 month after surgery (follow up visit)
  Adhesion: The primary end point will be assessed in terms of patient adhesion at the digital survey of the OKS index compared to the conventional one.
  Those who complete the questionnaire within 48 hours of the follow up visit will be considered as cases with positive adhesion with the digital assessment; those who reply after 48 hours or who do not reply will be considered with negative adhesion.
Patient's adhesion to the digital Oxford Knee Score compilation three months after surgery | 3 months after surgery (follow up visit)
  Adhesion: The primary end point will be assessed in terms of patient adhesion at the digital survey of the OKS index compared to the conventional one.
  Those who complete the questionnaire within 48 hours of the follow up visit will be considered as cases with positive adhesion with the digital assessment; those who reply after 48 hours or who do not reply will be considered with negative adhesion.
Patient's adhesion to the digital Oxfor Knee Score compilation six months after surgery | 6 months after surgery (follow up visit)
  Adhesion: The primary end point will be assessed in terms of patient adhesion at the digital survey of the OKS index compared to the conventional one.
  Those who complete the questionnaire within 48 hours of the follow up visit will be considered as cases with positive adhesion with the digital assessment; those who reply after 48 hours or who do not reply will be considered with negative adhesion.

SECONDARY OUTCOMES:
Level of coherence between the OKS detected on an outpatient basis by means of a paper questionnaire and that detected by digital extra-ambulatory administration one month before surgery | 1 month before surgery (pre-admission outpatient visit)
  As a secondary end point, the level of coherence between the Oxford Knee Score detected on an outpatient basis by means of a paper questionnaire and that detected by digital extra-ambulatory administration will be examined, one month before surgery, on the occasion of the pre-admission visit.
  Which and how many responses will be discordant with respect to the two types of survey will be indicated.
Level of coherence between the OKS detected on an outpatient basis by means of a paper questionnaire and that detected by digital extra-ambulatory administration one month after surgery | 1 month after surgery (follow up visit)
  As a secondary end point, the level of coherence between the Oxfor Knee Score detected on an outpatient basis by means of a paper questionnaire and that detected by digital extra-ambulatory administration will be examined, one month after surgery, on the occasion of the follow up visit.
  Which and how many responses will be discordant with respect to the two types of survey will be indicated.
Level of coherence between the OKS detected on an outpatient basis by means of a paper questionnaire and that detected by digital extra-ambulatory administration threee months after surgery | 3 months after surgery (follow up visit)
  As a secondary end point, the level of coherence between the Oxford Knee Score detected on an outpatient basis by means of a paper questionnaire and that detected by digital extra-ambulatory administration will be examined, three months after surgery, on the occasion of the follow up visit.
  Which and how many responses will be discordant with respect to the two types of survey will be indicated.
Level of coherence between the OKS detected on an outpatient basis by means of a paper questionnaire and that detected by digital extra-ambulatory administration six months after surgery | 6 months after surgery (follow up visit)
  As a secondary end point, the level of coherence between the Oxford Knee Score detected on an outpatient basis by means of a paper questionnaire and that detected by digital extra-ambulatory administration will be examined, six months after surgery, on the occasion of the follow up visit.
  Which and how many responses will be discordant with respect to the two types of survey will be indicated.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided